CLINICAL TRIAL: NCT06483542
Title: A Retrospective Analysis of the Impact of Non-nutritional Calories During Continuous Veno-Venous Hemofiltration
Brief Title: Bionenergetic Balance During CVVH
Acronym: BALANCE
Status: Active, not recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: BUN 1432022000231
Record Dates: First submitted 2023-01-24; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Acute Kidney Injury; Continuous Venovenous Hemofiltration; Energy Metabolism; Resting Energy Expenditure; Nutrition Therapy
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: all patients
  Interventions: Other: bioenergetic balance

INTERVENTIONS:
Other: bioenergetic balance — Bioenergetic balance is calculated for all patients who had a resting energy expenditure measurement with indirect calorimetry.

SUMMARY:
The bioenergetic balance is the sum of energy exchanged during CRRT and is mostly defined by citrate glucose and lactate. When CRRT was performed with the older dialysis fluids, glucose and lactate could be an important source of energy next to citrate when used as predilution (6, 7). During continuous venovenous hemofiltration (CVVH), a subgroup of CRRT which is performed with the newer dialysis fluids without lactate or glucose as advocated by the KDIGOguidelines, glucose and in a minor way lactate mostly induce a loss of energy. The first aim is to determine how this bioenergetic balance impacts energy need compared to the measured energy with indirect calorimetry and how nutrition therapy needs to be adapted.

Also, disease specific predicting equation have been created for patients suffering from acute kidney injury treated with renal replacement therapy. How this predicting equation and other existing predicting equations agree with the measured REE has not been validated yet. The second aim is to determine how predictive equations correlate with measured REE in patients treated with CVVH.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the adult ICU (01/01/2021-30/09/2022)
* At least one indirect calorimetry measurement (ventilator) or calculation based on harris benedict OR 25Kcal/kg/day
* Combined with bio energetic balance measurement
* Receiving CVVH during intensive care stay

Exclusion Criteria:

* Patients admitted outside of the inclusion period will be excluded
* The absence of an indirect calorimetry measurement (ventilator) or calculation - based on the Harris Benedict OR 25Kcal/kg/day formula OR The absence of a bio energetic balance measurement
* The absence of CVVH during intensive care stay
* Pediatric (intensive care unit) patients

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients with acute kidney injury who require CVVH
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Energy | during study completion, on average 4weeks
  expressed in Kcal

SECONDARY OUTCOMES:
resting energy expenditure | during study completion, on average 4weeks
  expressed in Kcal
protein to energy ratio | during study completion, on average 4weeks
  expressed in gr/Kcal

CONTACTS AND LOCATIONS:
Overall Officials: Joop Jonckheer, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair ziekenhuis Brussel, Jette, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
If IPD is asked for, anonymized raw data can be shared
Supporting Information: Study Protocol, CSR
Time Frame: From March 2023 until March 2053